CLINICAL TRIAL: NCT02340208
Title: A Phase I/II Open-Label, Non-Randomized Dose Escalation Study of Immunoconjugate L-DOS47 as a Monotherapy in Non-Squamous Non-Small Cell Lung Cancer Patients
Brief Title: A Phase I/II Open-Label, Non-Randomized Dose Escalation Study of Immunoconjugate L-DOS47
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Helix BioPharma Corporation (Industry)
Collaborators: Pharm-Olam International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LDOS002
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Neoplasms; Immunoconjugate; Tumor microenvironment alkalinization
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-DOS47 (Experimental): Patient will be recruited into cohorts of L-DOS47 escalating doses, with a minimum of 3 and a maximum of 6 patients per cohort. The starting dose of L-DOS47 will be 0.12 μg/kg; further possible dose levels include 0.21, 0.33, 0.46, 0.59, 0.78, 1.04, 1.38, 1.84, 2.45, 3.26 and 4.33 μg/kg.
  Interventions: Drug: L-DOS47

INTERVENTIONS:
Drug: L-DOS47 — A treatment cycle will be 21 days with patients receiving L-DOS47 on cycle Days 1 and 8.

SUMMARY:
The primary purpose of this research study is to evaluate how safe, how well tolerated and how effective a range of doses of L-DOS47 in patients with non-squamous non-small cell lung cancer when given as a monotherapy.

DETAILED DESCRIPTION:
Patients will be recruited into cohorts, with a minimum of three and a maximum of six patients per cohort. All patients at a given dose level must complete Cycle 1 (3 week period) before escalation in subsequent patients can proceed. The decision for dose escalation to the next dose level will be made after the safety and available pharmacokinetic (PK) data have been reviewed by the Trial Steering Committee (TSC).

Escalation of L-DOS47 will continue until a maximum tolerated dose (MTD) is reached.

After the MTD of L-DOS47 has been determined in Phase I, up to 20 patients will be enrolled (taken forward from Phase I) to evaluate the preliminary efficacy of L-DOS47 (i.e., response rate using the Response Evaluation Criteria in Solid Tumours [RECIST] version 1.1 criteria, disease progression and survival); monitoring will include radiologic evaluations every second cycle. The safety and tolerability of L-DOS47 will also be further evaluated. Pharmacokinetic information will be collected as well as relevant observations on the activity of L-DOS47.

For all patients, treatment with L-DOS47 will continue either until the patient experiences disease progression, unacceptable toxicity, the patient withdraws consent or has completed four treatment cycles and does not wish to continue with additional cycles, whichever occurs first. After four cycles, patients may continue to receive L-DOS47 for as long as there is sustained clinical benefit and it is well tolerated, in the opinion of the Investigator.

ELIGIBILITY:
Main Inclusion Criteria:

Patients will be entered in the study only if they meet all of the following criteria:

1. Male or female aged ≥ 18 years old
2. Have histologically confirmed non-squamous NSCLC that are:

   1. Chemo naïve Stage IIIb or IV non-squamous NSCLC who are not candidates for chemotherapy or radiotherapy, or who refused standard therapy
   2. Refractory Stage IIIb or IV non-squamous NSCLC. (Staging of non-squamous NSCLC must be assessed according to TNM, 7th edition and based on computed tomography (CT) scan.)
3. Have at least a single measurable lesion in accordance with the RECIST v1.1 criteria.
4. Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
5. Have a life expectancy of ≥ 3 months
6. Have adequate bone marrow, renal and liver function

Main Exclusion Criteria:

1. Are pregnant or nursing mother
2. Have a prior history of other malignancies with the exception of non melanoma skin cancer
3. Have known history of central nervous system (CNS) metastatic disease (previously treated or untreated)
4. Show evidence of active infection
5. Have received treatment in another clinical study within the 30 days before commencing study drug or have not recovered from side effects of a study drug, except for alopecia
6. Have a serious uncontrolled medical condition
7. Known positive human immunodeficiency virus (HIV), known hepatitis B surface antigen, or hepatitis C positive
8. Sustained QTc (QT interval corrected for heart rate) with Fridericia's correction > 450 ms at screening, or a history of additional risk factors for Torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome)
9. Pre-existing peripheral neuropathy ≥ CTC Grade 2
10. Have dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent or compliance with the requirements of the protocol
11. Are receiving chemotherapy during the 30 days before study treatment start; are receiving radiotherapy, targeted therapy, hormonal therapy, immunotherapy, major surgery or other study drugs during the 4 weeks before study treatment start, or have not recovered from all treatment related toxicities to Grade ≤ 1, except for alopecia. (Radiotherapy is allowed for the symptomatic treatment of bone metastases.)
12. Are taking systemic steroids (other than inhalers or topical steroids) or other medication to suppress the immune system
13. Are participating (or planning to participate) in any other clinical trial during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-05; Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of drug-related adverse events as a measure of safety and tolerability of L-DOS47 | Up to 12 weeks
  Assessed during the AE reporting period starts on Cycle 1 Day 1 up to the last study visit.

SECONDARY OUTCOMES:
L-DOS47 related toxicity during the first 2 hours after infusion | During the first 2 hours after infusion
  Assessed by the incidence and severity of AEs and SAEs and changes in vital signs
The incidence and severity of all reported adverse events and serious adverse events | Participants will be followed for 12 weeks and the 30 day follow-up period
  Assessed during the AE reporting period starts on Cycle 1 Day 1 up to the last study visit.
Changes from baseline for additional safety parameters (clinical laboratory assessments, vital signs, weight, oxygen requirement and 12-lead ECG) | Up to 12 weeks
  Safety parameters include clinical laboratory assessments, vital signs, weight, oxygen requirement and 12-lead ECG
The evaluation of anti-L-DOS47 antibody over time | Up to 12 weeks
  Serum samples will be collected and analyzed from all patients dosed with L-DOS47.

OTHER OUTCOMES:
Maximum observed plasma concentration (Cmax) of L-DOS47 at each dose level | Up to 12 weeks
  Pharmacokinetic parameters for L-DOS47 will be determined from plasma samples collected from all patient dosed with L-DOS47.
Time to maximum observed plasma concentration (Tmax) of L-DOS47 at each dose level | Up to 12 weeks
  Pharmacokinetic parameters for L-DOS47 will be determined from plasma samples collected from all patient dosed with L-DOS47.
Area under the concentration (AUC) vs time curve of L-DOS47 at each dose level | Up to 12 weeks
  Pharmacokinetic parameters for L-DOS47 will be determined from plasma samples collected from all patient dosed with L-DOS47.
Terminal elimination half-life of L-DOS47 at each dose level | Up to 12 weeks
  Pharmacokinetic parameters for L-DOS47 will be determined from plasma samples collected from all patient dosed with L-DOS47.

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Kowalski, MD, PhD, Principal Investigator — The Maria Sklodowska-Curie Memorial Cancer Centre & Institute of Oncology
Locations (5):
- Poland (5):
  - Mazovian Center of Pulmonary Diseases and Tuberculosis, Otwock
  - Med. Polonia Hospital Poznan, Poznan
  - Institute of Tuberculosis and Lung Diseases, Warsaw
  - Military Medical Institute, Warsaw
  - The Maria Sklodowska-Curie Memorial Cancer Centre & Institute of Oncology, Warsaw